CLINICAL TRIAL: NCT00729378
Title: Exercise and Bone Development in Young Girls
Brief Title: Jump-In: Building Better Bones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Scott Going, Department Head, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HD050775
Record Dates: First submitted 2008-08-05; First posted 2008-08-07 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2021-03

CONDITIONS: Adolescent Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Intervention (Experimental): Implementation of intervention program designed to provide skeletal loading through high impact activities. All activities performed by subjects in exercise intervention arm will be assessed by physical activity questionnaire and use of pedometer. Have baseline anthropometric measurements, total body DXA scans and peripheral quantitative computed tomography (pQCT) scans of the tibia and femur.
  Interventions: Other: Skeletal loading
- Control (No Intervention): Participants in this arm will not take part in exercise intervention. All activities performed by subjects in control arm will be assessed by physical activity questionnaire and use of pedometer. Have baseline anthropometric measurements, total body DXA scans and peripheral quantitative computed tomography (pQCT) scans of the tibia and femur.

INTERVENTIONS:
Other: Skeletal loading — Impact activities, 3 times per week, increasing the number of jumps (up to 40) and increasing height (from 6 inches to 24 inches per repetition) over the initial 8-weeks (2 months). New activities will be introduced approximately every 2-3 months in order to continually stress the skeleton over 2 years.
  Arms: Exercise Intervention

SUMMARY:
The Jump-In study will prospectively assess the effects of impact exercise on skeletal development in young girls, including bone mass, bone mineral density, and bone geometry. We hypothesize that girls who regularly participate in impact loading exercise will accrue greater skeletal mass, increase bone density and undergo structural adaptations that in combination will improve bone strength compared to girls who do not participate in impact exercise.

DETAILED DESCRIPTION:
Jump-In is a school-based, block-randomized, trial of the effects of impact-loading exercise on skeletal development in prepubescent and early pubescent girls. Fourth (n=~200) and sixth (n=~200) grade girls in 14 Tucson (Arizona) schools with no contraindication to physical exercise will be enrolled. Girls in intervention schools will participate in impact activities 3 times per week at school, progressively increasing the number (up to 40) of jumps and their height (from 6 inches to 18 inches per repetition) over the initial 2 months. Thereafter, new activities will be introduced approximately every 2-3 months to maintain interest and motivation, and continually stress the skeleton in novel ways, over 2 years of intervention. Physical and behavioral assessments will be done in both intervention and control groups at baseline, end of the initial school year, and yearly thereafter for 5 years. Assessments include height and weight, selected skeletal lengths, fat, lean soft tissue, bone mineral content and areal density from dual energy x-ray absorptiometry (DXA), and bone geometry (e.g., cortical thickness, periosteal circumference and cortical and trabecular density) and muscle area from peripheral quantitative computed tomography (pQCT). Also, maturation will be assessed via the Tanner Stage (self-assessment against standardized drawings of stages of physical development), diet from the Harvard Youth Food Frequency Questionnaire, and physical activity using pedometers and standardized questionnaires. We hypothesize that girls in intervention schools will demonstrate enhanced skeletal development, including greater mineral mass and density, and enhanced bone geometry, leading to greater bone strength compared to girls in control schools. We further hypothesize that younger (Tanner Stage 1) girls will experience greater adaptations than older girls (Tanner 2 and 3), and that positive adaptations will be maintained throughout the 3-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

female; entering 4th or 6th grade at enrollment; and willing and able to undergo all of the testing requirements; no physical conditions that limit participation in physical activity/exercise; able to read and write English.

Exclusion Criteria:

Girls with severe learning disabilities (identified by schools), who are unable to complete questionnaires or otherwise comply with assessment protocols will be excluded. Any subjects (or potential subjects) suffering from medical conditions and/or disabilities that would limit their participation in exercise will be excluded from the study, following the American Academy of Pediatrics (AAP) guidelines. Further, any volunteers who are taking medications that would limit exercise and/or alter bone mineral accrual will also be excluded from the study. Girls with a positive pregnancy screening test at the time of the lab visit before DXA scanning will be excluded.

Ages: 9 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 509 (Actual)
Dates: Start 2007-04; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Going, Ph.D., Principal Investigator — University of Arizona-Dept. of Nutritional Sciences
Locations (1):
- University of Arizona-Ina Gittings Bldg. #93, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farr JN, Van Loan MD, Lohman TG, Going SB. Lower physical activity is associated with skeletal muscle fat content in girls. Med Sci Sports Exerc. 2012 Jul;44(7):1375-81. doi: 10.1249/MSS.0b013e31824749b2. PMID 22217562
- [Derived] Farr JN, Tomas R, Chen Z, Lisse JR, Lohman TG, Going SB. Lower trabecular volumetric BMD at metaphyseal regions of weight-bearing bones is associated with prior fracture in young girls. J Bone Miner Res. 2011 Feb;26(2):380-7. doi: 10.1002/jbmr.218. PMID 20721933

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed for three years (2007-2009) in a total of 16 elementary and middle schools (9 intervention and 7 control) in two Tucson, Arizona area school districts. Recruitment consisted of attending back to school days and holding recruitment assemblies before or after school.
Pre-assignment Details: Intervention and control schools designated prior to recruiting. Schools were selected based on size, demographics, and student flow from elementary to middle school to prevent contamination. 739 participants completed informed consent process (agreed to participate); only 509 scheduled measurement appointments and completed study measurements.
Groups:
- Exercise Intervention: Subjects in the exercise intervention arm performed activities designed to provide skeletal loading: impact activities, 3 times per week, increasing the number of jumps (up to 40) and increasing height (from 6 inches to 24 inches per repetition) over the initial 8-weeks (2 months). New activities were introduced approximately every 2-3 months in order to continually stress the skeleton over 2 years.
  Physical activity performed by these subjects (in addition to intervention activities) was objectively assessed by pedometer (7-day wear period) and further assessed by a validated past year physical activity questionnaire PYPAQ).
- Control: Subjects in the control arm did not take part in intervention exercises. Physical activity performed by these subjects was objectively assessed by pedometer (7-day wear period) and further assessed by a validated past year physical activity questionnaire PYPAQ).
Period: Baseline
Arm/Group | Exercise Intervention | Control
Started | 430 | 309
Completed | 292 | 217
Not Completed | 138 | 92
Not completed — Did not complete study measurements | 72 | 33
Not completed — Withdrawal by Subject | 66 | 59
Period: 12-months
Arm/Group | Exercise Intervention | Control
Started | 292 | 217
Completed | 192 | 152
Not Completed | 100 | 65
Not completed — Lost to Follow-up | 100 | 65
Period: 24-months
Arm/Group | Exercise Intervention | Control
Started | 192 | 152
Completed | 120 | 101
Not Completed | 72 | 51
Not completed — Lost to Follow-up | 72 | 51
Period: 36-months
Arm/Group | Exercise Intervention | Control
Started | 120 | 101
Completed | 105 | 95
Not Completed | 15 | 6
Not completed — Lost to Follow-up | 15 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Intervention | Control | Total
Number analyzed (Participants) | 292 | 217 | 509
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (1.1) | 10.7 (1.0) | 10.7 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 292 | 217 | 509
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67 | 50 | 117
  Not Hispanic or Latino | 225 | 167 | 392
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 20 | 11 | 31
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 11 | 3 | 14
  White | 254 | 196 | 450
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 292 | 217 | 509

OUTCOME MEASURES:

1. Primary Outcome: Baseline Total Volumetric Bone Density at the Femur 4% Site
Description: Baseline (initial) measurement of total volumetric bone density at the femur 4% site. Measurement made by peripheral quantitative computed tomography (pQCT) at a distance of 4% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: Population consists of all participants that had complete measurements at the baseline time point (N = 503; Age = 10.6 +/- 1.1 yrs; Height = 144.5 +/- 9.7 cm; Weight = 39.2 +/- 10.5 kg).
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Groups:
- Exercise Intervention: Participants randomized to the exercise intervention group performed activities designed to provide skeletal loading: impact activities 3 times per week, increasing the number of jumps (up to 40) and increasing height (from 6 inches to 24 inches per repetition) over the initial 8-weeks (2 months). New activities were introduced approximately every 2-3 months in order to continually stress the skeleton over 2 years.
  Physical activity performed by these subjects (in addition to intervention activities) was objectively assessed by pedometer (7-day wear period) and further assessed by a validated past year physical activity questionnaire PYPAQ).
- Control: Participants randomized to the control arm did not perform intervention activities. Physical activity was objectively assessed by pedometer (7-day wear period) and further assessed by a validated past year physical activity questionnaire (PYPAQ).
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 277.25 (33.83) | 270.79 (32.97)

2. Primary Outcome: Baseline Volumetric Bone Density of Trabecular Bone at the Femur 4% Site
Description: Baseline (initial) measurement of volumetric bone density of trabecular bone at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 239.32 (32.2) | 232.34 (31.56)

3. Primary Outcome: Baseline Volumetric Bone Density of Cortical Bone at the Femur 4% Site
Description: Baseline (initial) measurement of volumetric bone density of Cortical bone at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 273.80 (31.23) | 267.89 (30.75)

4. Primary Outcome: Baseline Trabecular Bone Area at the Femur 4% Site
Description: Baseline (initial) measurement of trabecular bone area at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: square millimeters (mm^2).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
millimeters squared (mm^2) | 1039.55 (220.17) | 1053.15 (227.32)

5. Primary Outcome: Baseline Cortical Bone Area at the Femur 4% Site
Description: Baseline (initial) measurement of cortical bone area at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: square millimeters (mm^2).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
millimeters squared (mm^2) | 1335.56 (274.22) | 1348.65 (284.24)

6. Primary Outcome: Baseline Periosteal Circumference at the Femur 4% Site
Description: Baseline (initial) measurement of periosteal circumference at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
millimeters (mm) | 124.91 (12.42) | 125.63 (12.50)

7. Primary Outcome: Baseline Bone Strength Index at the Femur 4% Site
Description: Baseline (initial) measurement of bone strength index (BSI) at the femur 4% site. Bone Strength Index (BSI) is a measurement of the resistance to compression forces at the epiphyses of long bones. Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: mm^4.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^4
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
mm^4 | 96.77 (28.00) | 93.52 (27.39)

8. Primary Outcome: Baseline Total Volumetric Bone Density at the Femur 20% Site
Description: Baseline (initial) measurement of total volumetric bone density at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 489.70 (63.98) | 478.72 (60.59)

9. Primary Outcome: Baseline Volumetric Bone Density of Trabecular Bone at the Femur 20% Site
Description: Baseline (initial) measurement of volumetric bone density of trabecular bone at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 163.81 (39.43) | 153.11 (36.77)

10. Primary Outcome: Baseline Volumetric Bone Density of Cortical Bone at the Femur 20% Site
Description: Baseline (initial) measurement of volumetric bone density of Cortical bone at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 1046.01 (22.27) | 1045.20 (23.07)

11. Primary Outcome: Baseline Periosteal Circumference at the Femur 20% Site
Description: Baseline (initial) measurement of periosteal circumference at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
millimeters (mm) | 77.43 (8.56) | 77.78 (8.66)

12. Primary Outcome: Baseline Cortical Thickness at the Femur 20% Site
Description: Baseline (initial) measurement of cortical thickness at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
millimeters (mm) | 2.52 (.37) | 2.50 (.35)

13. Primary Outcome: Baseline Stress-Strain Index at the Femur 20% Site
Description: Baseline (initial) measurement of stress-strain index at the femur 20% site. Stress-strain index (also called strength-strain index and stress-strength index in the literature) is a measure of the resistance to torsional and bending forces at diaphyseal sites of long bones. Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: mm^3.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
mm^3 | 1340.19 (404.78) | 1344.66 (399.31)

14. Primary Outcome: Baseline Volumetric Bone Density of Trabecular Bone at the Tibia 4% Site
Description: Baseline (initial) measurement of volumetric bone density of trabecular bone at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 224.03 (27.58) | 219.74 (25.56)

15. Primary Outcome: Baseline Total Volumetric Bone Density at the Tibia 4% Site
Description: Baseline (initial) measurement of total volumetric bone density at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 297.27 (37.02) | 291.62 (33.17)

16. Primary Outcome: Baseline Volumetric Bone Density of Cortical Bone at the Tibia 4% Site
Description: Baseline (initial) measurement of volumetric bone density of cortical bone at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 297.40 (35.63) | 291.93 (31.92)

17. Primary Outcome: Baseline Trabecular Bone Area at the Tibia 4% Site
Description: Baseline (initial) measurement of trabecular bone area at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: square millimeters (mm^2).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
millimeters squared (mm^2) | 467.73 (100.86) | 475.80 (108.85)

18. Primary Outcome: Baseline Cortical Bone Area at the Tibia 4% Site
Description: Baseline (initial) measurement of cortical bone area at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: square millimeters (mm^2).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
millimeters squared (mm^2) | 617.19 (117.67) | 625.57 (127.11)

19. Primary Outcome: Baseline Periosteal Circumference at the Tibia 4% Site
Description: Baseline (initial) measurement of periosteal circumference at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
millimeters (mm) | 85.86 (8.36) | 86.43 (8.82)

20. Primary Outcome: Baseline Bone Strength Index at the Tibia 4% Site
Description: Baseline (initial) measurement of bone strength index (BSI) at the tibia 4% site. Bone Strength Index (BSI) is a measurement of the resistance to compression forces at the epiphyses of long bones. Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: mm^4.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^4
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
mm^4 | 52.45 (15.15) | 51.03 (13.63)

21. Primary Outcome: Baseline Total Volumetric Bone Density at the Tibia 50% Site
Description: Baseline (initial) measurement of total volumetric bone density at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 745.69 (59.54) | 736.33 (58.07)

22. Primary Outcome: Baseline Volumetric Bone Density of Trabecular Bone at the Tibia 50% Site
Description: Baseline (initial) measurement of volumetric bone density of trabecular bone at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 137.39 (26.83) | 131.63 (26.97)

23. Primary Outcome: Baseline Volumetric Bone Density of Cortical Bone at the Tibia 50% Site
Description: Baseline (initial) measurement of volumetric bone density of cortical bone at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 1070.32 (32.88) | 1070.95 (31.93)

24. Primary Outcome: Baseline Periosteal Circumference at the Tibia 50% Site
Description: Baseline (initial) measurement of periosteal circumference at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
millimeters (mm) | 61.98 (5.43) | 62.33 (5.83)

25. Primary Outcome: Baseline Cortical Thickness at the Tibia 50% Site
Description: Baseline (initial) measurement of cortical thickness at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
millimeters (mm) | 4.05 (.58) | 4.00 (.54)

26. Primary Outcome: Baseline Stress-Strain Index at the Tibia 50% Site
Description: Baseline (initial) measurement of stress-strain index at the tibia 50% site. Stress-strain index (also called strength-strain index and stress-strength index in the literature) is a measure of the resistance to torsional and bending forces at diaphyseal sites of long bones. Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: mm^3.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
mm^3 | 1004.97 (272.40) | 1023.74 (297.42)

27. Primary Outcome: Baseline Total Volumetric Bone Density at the Tibia 66% Site
Description: Baseline (initial) measurement of total volumetric bone density at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 566.04 (63.11) | 552.71 (61.05)

28. Primary Outcome: Baseline Volumetric Bone Density of Trabecular Bone at the Tibia 66% Site
Description: Baseline (initial) measurement of volumetric bone density of trabecular bone at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 159.04 (30.48) | 152.34 (28.73)

29. Primary Outcome: Baseline Volumetric Bone Density of Cortical Bone at the Tibia 66% Site
Description: Baseline (initial) measurement of volumetric bone density of cortical bone at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
milligrams per cubic centimeter (mg/ccm) | 1029.42 (32.92) | 1026.07 (31.38)

30. Primary Outcome: Baseline Periosteal Circumference at the Tibia 66% Site
Description: Baseline (initial) measurement of periosteal circumference at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
millimeters (mm) | 71.55 (6.53) | 72.34 (7.25)

31. Primary Outcome: Baseline Cortical Thickness at the Tibia 66% Site
Description: Baseline (initial) measurement of cortical thickness at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
millimeters (mm) | 3.06 (.49) | 3.02 (.46)

32. Primary Outcome: Baseline Stress-Strain Index at the Tibia 66% Site
Description: Baseline (initial) measurement of strength-strain index at the tibia 66% site. Stress-strain index (also called strength-strain index and stress-strength index in the literature) is a measure of the resistance to torsional and bending forces at diaphyseal sites of long bones. Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: mm^3.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 286 | 217
mm^3 | 1167.94 (331.61) | 1187.31 (353.09)

33. Primary Outcome: 12-month Change in Total Volumetric Bone Density the Femur 4% Site
Description: Baseline to 12-month change in total volumetric bone density at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: Population consists of all participants that had complete measurements at the baseline, 12-month and 24-month time points (N=207). At 12-months: Age=11.8 +/- 1.0 yrs; Height=153.3 +/- 9.9 cm; Weight=44.0 +/- 9.3 kg. At 24-months: Age=12.8 +/- 1.0 yrs; Height=158.8 +/- 9.1 cm; Weight=50.0 +/- 10.7 kg.
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Groups:
- Exercise Intervention Group: Participants randomized to the exercise intervention group performed activities designed to provide skeletal loading: impact activities 3 times per week, increasing the number of jumps (up to 40) and increasing height (from 6 inches to 24 inches per repetition) over the initial 8-weeks (2 months). New activities were introduced approximately every 2-3 months in order to continually stress the skeleton over 2 years.
  Physical activity performed by these subjects (in addition to intervention activities) was objectively assessed by pedometer (7-day wear period) and further assessed by a validated past year physical activity questionnaire PYPAQ).
- Control Group: Participants randomized to the control arm did not perform intervention activities. Physical activity was objectively assessed by pedometer (7-day wear period) and further assessed by a validated past year physical activity questionnaire (PYPAQ).
Arm/Group | Exercise Intervention Group | Control Group
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 3.10 (15.36) | 2.83 (12.32)

34. Primary Outcome: 12-month Change in Volumetric Bone Density of Trabecular Bone at the Femur 4% Site
Description: Baseline to 12-month change in volumetric bone density of trabecular bone at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention Group | Control Group
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 3.37 (15.23) | 5.89 (12.94)

35. Primary Outcome: 12-month Change in Volumetric Bone Density of Cortical Bone at the Femur 4% Site
Description: Baseline to 12-month change in volumetric bone density of cortical bone at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention Group | Control Group
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 2.14 (14.47) | 1.68 (11.47)

36. Primary Outcome: 12-month Change in Trabecular Bone Area at the Femur 4% Site
Description: Baseline to 12-month change in trabecular bone area at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: square millimeters (mm^2).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters squared (mm^2) | 104.16 (111.80) | 144.97 (96.38)

37. Primary Outcome: 12-month Change in Cortical Bone Area at the Femur 4% Site
Description: Baseline to 12-month change in cortical bone area at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: square millimeters (mm^2).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters squared (mm^2) | 140.00 (131.17) | 185.50 (119.42)

38. Primary Outcome: 12-month Change in Periosteal Circumference at the Femur 4% Site
Description: Baseline to 12-month change in periosteal circumference at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | 6.17 (5.80) | 8.09 (4.84)

39. Primary Outcome: 12-month Change in Bone Strength Index at the Femur 4% Site
Description: Baseline to 12-month change in bone strength index (BSI) at the femur 4% site. Bone Strength Index (BSI) is a measurement of the resistance to compression forces at the epiphyses of long bones. Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: mm^4.
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mm^4
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
mm^4 | 12.84 (12.67) | 15.03 (14.19)

40. Primary Outcome: 12-month Change in Total Volumetric Bone Density at the Femur 20% Site
Description: Baseline to 12-month change in total volumetric bone density at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 2.40 (22.38) | -2.46 (18.74)

41. Primary Outcome: 12-month Change in Volumetric Bone Density of Trabecular Bone at the Femur 20% Site
Description: Baseline to 12-month change in volumetric bone density of trabecular bone at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 7.12 (12.98) | 5.77 (12.38)

42. Primary Outcome: 12-month Change in Volumetric Bone Density of Cortical Bone at the Femur 20% Site
Description: Baseline to 12-month change in volumetric bone density of cortical bone at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 6.87 (20.02) | 4.39 (19.38)

43. Primary Outcome: 12-month Change in Thickness of Cortical Bone at the Femur 20% Site
Description: Baseline to 12-month change in thickness of cortical bone at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units millimeters (mm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | .11 (.17) | .11 (.15)

44. Primary Outcome: 12-month Change in Periosteal Circumference at the Femur 20% Site
Description: Baseline to 12-month change in periosteal circumference at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | 4.89 (2.21) | 5.65 (2.20)

45. Primary Outcome: 12-month Change in Stress-Strain Index at the Femur 20% Site
Description: Baseline to 12-month change in strength-strain index at the femur 20% site. Stress-strain index (also called strength-strain index and stress-strength index in the literature) is a measure of the resistance to torsional and bending forces at diaphyseal sites of long bones. Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: mm^3.
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
mm^3 | 261.94 (137.73) | 297.43 (145.31)

46. Primary Outcome: 12-month Change in Total Volumetric Bone Density at the Tibia 4% Site
Description: Baseline to 12-month change in total volumetric bone density at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 9.87 (17.29) | 10.34 (19.34)

47. Primary Outcome: 12-month Change in Volumetric Bone Density of Trabecular Bone at the Tibia 4% Site
Description: Baseline to 12-month change in volumetric bone density of trabecular bone at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 2.84 (10.22) | 2.36 (9.33)

48. Primary Outcome: 12-month Change in Volumetric Bone Density of Cortical Bone at the Tibia 4% Site
Description: Baseline to 12-month change in volumetric bone density of cortical bone at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 9.69 (16.76) | 10.10 (18.73)

49. Primary Outcome: 12-month Change in Trabecular Bone Area at the Tibia 4% Site
Description: Baseline to 12-month change in trabecular bone area at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: square millimeters (mm^2).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters squared (mm^2) | 29.87 (52.91) | 24.65 (50.00)

50. Primary Outcome: 12-month Change in Cortical Bone Area at the Tibia 4% Site
Description: Baseline to 12-month change in cortical bone area at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: square millimeters (mm^2).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters squared (mm^2) | 44.85 (54.14) | 39.53 (49.12)

51. Primary Outcome: 12-month Change in Periosteal Circumference at the Tibia 4% Site
Description: Baseline to 12-month change in periosteal circumference at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | 3.17 (3.70) | 2.77 (3.44)

52. Primary Outcome: 12-month Change in Bone Strength Index at the Tibia 4% Site
Description: Baseline to 12-month change in bone strength index (BSI) at the tibia 4% site. Bone Strength Index (BSI) is a measurement of the resistance to compression forces at the epiphyses of long bones. Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: mm^4.
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mm^4
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
mm^4 | 7.84 (5.39) | 7.46 (5.53)

53. Primary Outcome: 12-month Change in Total Volumetric Bone Density at the Tibia 50% Site
Description: Baseline to 12-month change in total volumetric bone density at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 17.98 (22.27) | 17.76 (22.02)

54. Primary Outcome: 12-month Change in Volumetric Bone Density of Trabecular Bone at the Tibia 50% Site
Description: Baseline to 12-month change in volumetric bone density of trabecular bone at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | -2.74 (13.55) | -3.16 (15.63)

55. Primary Outcome: 12-month Change in Volumetric Bone Density of Cortical Bone at the Tibia 50% Site
Description: Baseline to 12-month change in volumetric bone density of cortical bone at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 14.34 (22.23) | 11.16 (18.91)

56. Primary Outcome: 12-month Change in Periosteal Circumference at the Tibia 50% Site
Description: Baseline to 12-month change in periosteal circumference at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | 2.98 (1.33) | 3.11 (1.09)

57. Primary Outcome: 12-month Change in Cortical Thickness at the Tibia 50% Site
Description: Baseline to 12-month change in cortical thickness at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | .29 (.20) | .31 (.20)

58. Primary Outcome: 12-month Change in Stress-Strain Index at the Tibia 50% Site
Description: Baseline to 12-month change in strength-strain index at the tibia 50% site. Stress-strain index (also called strength-strain index and stress-strength index in the literature) is a measure of the resistance to torsional and bending forces at diaphyseal sites of long bones. Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: mm^3.
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
mm^3 | 171.82 (68.00) | 185.36 (79.04)

59. Primary Outcome: 12-month Change in Total Volumetric Bone Density at the Tibia 66% Site
Description: Baseline to 12-month change in total volumetric bone density at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 7.00 (32.41) | 9.58 (29.98)

60. Primary Outcome: 12-month Change in Volumetric Bone Density of Trabecular Bone at the Tibia 66% Site
Description: Baseline to 12-month change in volumetric bone density of trabecular bone at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate.Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 3.40 (13.49) | 2.08 (14.64)

61. Primary Outcome: 12-month Change in Volumetric Bone Density of Cortical Bone at the Tibia 66% Site
Description: Baseline to 12-month change in volumetric bone density of cortical bone at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 9
milligrams per cubic centimeter (mg/ccm) | 11.63 (24.00) | 12.69 (21.32)

62. Primary Outcome: 12-month Change in Periosteal Circumference at the Tibia 66% Site
Description: Baseline to 12-month change in periosteal circumference at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | 3.69 (2.35) | 3.79 (2.06)

63. Primary Outcome: 12-month Change in Cortical Thickness at the Tibia 66% Site
Description: Baseline to 12-month change in cortical thickness at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | .17 (.21) | .18 (.22)

64. Primary Outcome: 12-month Change in Stress-Strain Index at the Tibia 66% Site
Description: Baseline to 12-month change in strength-strain index at the tibia 66% site. Stress-strain index (also called strength-strain index and stress-strength index in the literature) is a measure of the resistance to torsional and bending forces at diaphyseal sites of long bones. Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: mm^3.
Time Frame: Baseline to 12-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
mm^3 | 214.93 (96.58) | 228.46 (103.48)

65. Primary Outcome: 24-month in Change in Total Volumetric Bone Density the Femur 4% Site
Description: Baseline to 24-month change in total volumetric bone density at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units mg/ccm.
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention Group | Control Group
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 13.70 (22.89) | 13.47 (19.09)

66. Primary Outcome: 24-month in Change in Volumetric Bone Density of Trabecular Bone at the Femur 4% Site
Description: Baseline to 24-month change in volumetric bone density of trabecular bone at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention Group | Control Group
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 8.03 (19.34) | 8.23 (16.35)

67. Primary Outcome: 24-month in Change in Volumetric Bone Density of Cortical Bone at the Femur 4% Site
Description: Baseline to 24-month change in volumetric bone density of cortical bone at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention Group | Control Group
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 10.67 (21.83) | 10.78 (17.95)

68. Primary Outcome: 24-month Change in Trabecular Bone Area at the Femur 4% Site
Description: Baseline to 24-month change in trabecular bone area at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: square millimeters (mm^2).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Groups:
- Exercise Intervention: Participants randomized to the exercise intervention group performed activities designed to provide skeletal loading: impact activities 3 times per week, increasing the number of jumps (up to 40) and increasing height (from 6 inches to 24 inches per repetition) over the initial 8-weeks (2 months). New activities were introduced approximately every 2-3 months in order to continually stress the skeleton over 2 years.
  Physical activity performed by these subjects (in addition to intervention activities) was objectively assessed by pedometer (7-day wear period) and further assessed by a validated past year physical activity questionnaire PYPAQ).
  .
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters squared (mm^2) | 160.89 (158.53) | 178.04 (146.00)

69. Primary Outcome: 24-month Change in Cortical Bone Area at the Femur 4% Site
Description: Baseline to 24-month change in cortical bone area at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: square millimeters (mm^2).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters squared (mm^2) | 237.12 (178.61) | 255.67 (165.23)

70. Primary Outcome: 24-month Change in Periosteal Circumference at the Femur 4% Site
Description: Baseline to 24-month change in periosteal circumference at the femur 4% site . Measurement made by pQCT at a distance of 4% of total femur length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | 10.08 (7.73) | 10.72 (6.88)

71. Primary Outcome: 24-month Change in Bone Strength Index at the Femur 4% Site
Description: Baseline to 24-month change in bone strength index (BSI) at the femur 4% site. Bone Strength Index (BSI) is a measurement of the resistance to compression forces at the epiphyses of long bones. Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: mm^4.
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mm^4
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
mm^4 | 28.08 (17.51) | 27.81 (17.76)

72. Primary Outcome: 24-month Change in Total Volumetric Bone Density at the Femur 20% Site
Description: Baseline to 24-month change in total volumetric bone density at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 14.88 (31.73) | 15.36 (28.47)

73. Primary Outcome: 24-month Change in Volumetric Bone Density of Trabecular Bone at the Femur 20% Site
Description: Baseline to 24-month change in volumetric bone density of trabecular bone at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 11.83 (17.20) | 9.04 (13.87)

74. Primary Outcome: 24-month Change in Volumetric Bone Density of Cortical Bone at the Femur 20% Site
Description: Baseline to 24-month change in volumetric bone density of cortical bone at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 21.56 (29.46) | 22.26 (29.62)

75. Primary Outcome: 24-month Change in Thickness of Cortical Bone at the Femur 20% Site
Description: Baseline to 24-month change in thickness of cortical bone at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | .27 (.22) | .31 (.21)

76. Primary Outcome: 24-month Change in Periosteal Circumference at the Femur 20% Site
Description: Baseline to 24-month change in periosteal circumference at the femur 20% site . Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | 8.25 (3.38) | 9.29 (3.08)

77. Primary Outcome: 24-month Change in Stress-Strain Index at the Femur 20% Site
Description: Baseline to 24-month change in strength-strain index at the femur 20% site. Stress-strain index (also called strength-strain index and stress-strength index in the literature) is a measure of the resistance to torsional and bending forces at diaphyseal sites of long bones. Measurement made by pQCT at a distance of 20% of total femur length from the distal growth plate. Measurement units: mm^3.
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
mm^3 | 504.12 (202.34) | 582.69 (202.42)

78. Primary Outcome: 24-month Change in Total Volumetric Bone Density at the Tibia 4% Site
Description: Baseline to 24-month change in total volumetric bone density at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 28.22 (30.58) | 26.76 (29.35)

79. Primary Outcome: 24-month Change in Volumetric Bone Density of Trabecular Bone at the Tibia 4% Site
Description: Baseline to 24-month change in volumetric bone density of trabecular bone at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 7.37 (13.97) | 7.23 (17.18)

80. Primary Outcome: 24-month Change in Volumetric Bone Density of Cortical Bone at the Tibia 4% Site
Description: Baseline to 24-month change in volumetric bone density of cortical bone at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 27.29 (29.54) | 25.94 (28.46)

81. Primary Outcome: 24-month Change in Trabecular Bone Area at the Tibia 4% Site
Description: Baseline to 24-month change in trabecular bone area at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: square millimeters (mm^2).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters squared (mm^2) | 34.81 (70.70) | 35.83 (75.98)

82. Primary Outcome: 24-month Change in Cortical Bone Area at the Tibia 4% Site
Description: Baseline to 24-month change in cortical bone area at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: square millimeters (mm^2).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters squared (mm^2) | 65.50 (69.84) | 66.42 (73.94)

83. Primary Outcome: 24-month Change in Periosteal Circumference at the Tibia 4% Site
Description: Baseline to 24-month change in periosteal circumference at the tibia 4% site . Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | 4.64 (4.82) | 4.65 (5.15)

84. Primary Outcome: 24-month Change in Bone Strength Index at the Tibia 4% Site
Description: Baseline to 24-month change in bone strength index (BSI) at the tibia 4% site. Bone Strength Index (BSI) is a measurement of the resistance to compression forces at the epiphyses of long bones. Measurement made by pQCT at a distance of 4% of total tibia length from the distal growth plate. Measurement units: mm^4.
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mm^4
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
mm^4 | 17.28 (9.35) | 16.86 (10.14)

85. Primary Outcome: 24-month Change in Total Volumetric Bone Density at the Tibia 50% Site
Description: Baseline to 24-month change in total volumetric bone density at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 37.26 (29.74) | 39.83 (32.94)

86. Primary Outcome: 24-month Change in Volumetric Bone Density of Trabecular Bone at the Tibia 50% Site
Description: Baseline to 24-month change in volumetric bone density of trabecular bone at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | -3.51 (15.84) | -4.00 (14.16)

87. Primary Outcome: 24-month Change in Volumetric Bone Density of Cortical Bone at the Tibia 50% Site
Description: Baseline to 24-month change in volumetric bone density of cortical bone at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 33.70 (27.35) | 31.06 (26.75)

88. Primary Outcome: 24-month Change in Periosteal Circumference at the Tibia 50% Site
Description: Baseline to 24-month measurement of periosteal circumference at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | 5.26 (2.12) | 5.27 (1.63)

89. Primary Outcome: 24-month Change in Cortical Thickness at the Tibia 50% Site
Description: Baseline to 24-month change in cortical thickness at the tibia 50% site . Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | .51 (.28) | .53 (.28)

90. Primary Outcome: 24-month Change in Stress-Strain Index at the Tibia 50% Site
Description: Baseline to 24-month change in strength-strain index at the tibia 50% site. Stress-strain index (also called strength-strain index and stress-strength index in the literature) is a measure of the resistance to torsional and bending forces at diaphyseal sites of long bones. Measurement made by pQCT at a distance of 50% of total tibia length from the distal growth plate. Measurement units: mm^3.
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
mm^3 | 322.78 (114.10) | 336.49 (112.47)

91. Primary Outcome: 24-month Change in Total Volumetric Bone Density at the Tibia 66% Site
Description: Baseline to 24-month change in total volumetric bone density at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 17.83 (38.18) | 19.26 (41.46)

92. Primary Outcome: 24-month Change in Volumetric Bone Density of Trabecular Bone at the Tibia 66% Site
Description: Baseline to 24-month change in volumetric bone density of trabecular bone at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 4.48 (14.20) | 1.69 (16.02)

93. Primary Outcome: 24-month Change in Volumetric Bone Density of Cortical Bone at the Tibia 66% Site
Description: Baseline to 24-month change in volumetric bone density of cortical bone at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: milligrams per cubic centimeter (mg/ccm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter (mg/ccm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
milligrams per cubic centimeter (mg/ccm) | 28.96 (28.71) | 31.06 (28.49)

94. Primary Outcome: 24-month Change in Periosteal Circumference at the Tibia 66% Site
Description: Baseline to 24-month change in periosteal circumference at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | 6.75 (3.07) | 6.82 (3.06)

95. Primary Outcome: 24-month Change in Cortical Thickness at the Tibia 66% Site
Description: Baseline to 24-month change in cortical thickness at the tibia 66% site . Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: millimeters (mm).
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
millimeters (mm) | .32 (.27) | .32 (.31)

96. Primary Outcome: 24-month Change in Stress-Strain Index at the Tibia 66% Site
Description: Baseline to 24-month change in strength-strain index at the tibia 66% site. Stress-strain index (also called strength-strain index and stress-strength index in the literature) is a measure of the resistance to torsional and bending forces at diaphyseal sites of long bones. Measurement made by pQCT at a distance of 66% of total tibia length from the distal growth plate. Measurement units: mm^3.
Time Frame: Baseline to 24-months
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Exercise Intervention | Control
Number analyzed (Participants) | 109 | 98
mm^3 | 421.49 (172.67) | 435.13 (164.78)

ADVERSE EVENTS:
Time Frame: Since the time frame was based on a "school year", adverse event data were collected twice a year (at the end of each school semester) for up to 5 years (the duration of the study).
Groups:
- Exercise Intervention Arm: Implementation of intervention program designed to provide skeletal loading through high impact activities.
  Skeletal loading: impact activities, 3 times per week, increasing the number of jumps (up to 40) and increasing height (from 6 inches to 24 inches per repetition) over the initial 8-weeks (2 months). New activities will be introduced approximately every 2-3 months in order to continually stress the skeleton over 2 years.
- Control Arm: Participants in this arm will not take part in intervention exercises. All activities performed by subjects in control arm will be assessed by physical activity questionnaire and use of pedometer.
Arm/Group | Exercise Intervention Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/292 | 0/217
Other Adverse Events (participants affected / at risk) | 0/292 | 0/217

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes